CLINICAL TRIAL: NCT04667494
Title: Ultrasound Therapy In Cardiac Amyloidosis
Acronym: UTICA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sharmila Dorbala, Director, Nuclear Cardiology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003179
Record Dates: First submitted 2020-12-03; First posted 2020-12-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Amyloidosis Cardiac
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Intervention Model Description: Outcome measures will be evaluated before and after intervention with sonotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Sonotherapy (Experimental): All participants will undergo sonotherapy
  Interventions: Combination Product: Sonotherapy

INTERVENTIONS:
Combination Product: Sonotherapy — Use of high mechanical index ultrasound therapy with intravenous Definity contrast infusion

SUMMARY:
This is a prospective pilot clinical study of subjects with cardiac amyloidosis and control subjects without amyloidosis where we plan to evaluate changes in myocardial blood flow, systolic and diastolic function before and after sonotherapy.

DETAILED DESCRIPTION:
70 subjects will be enrolled in this study in 3 study groups: A) 30 subjects with light chain cardiac amyloidosis B) 30 subjects with transthyretin cardiac amyloidosis and C) 10 subjects without amyloidosis. All subjects will undergo rest 2D echocardiography, rest N-13 ammonia or rubidium-82 perfusion PET, Definity infusion with high mechanical index (MI) imaging defined as sonotherapy in this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years for AL-CA, > 65 years for ATTR-CA, > 65 years for controls
* Willing and able to provide consent
* Diagnosis of systemic light chain amyloidosis by standard criteria (see below) and in hematological remission (normal serum free light chain levels)

  * (immunofixation of serum and urine, IgG free light chain (FLC) assay, a biopsy of fat pad/ bone marrow, or organ biopsy, followed by typing of the light chain using immunohistochemistry or immunogold assay with confirmation by Mass spectroscopy as needed) AND
  * proof of cardiac involvement by AL amyloidosis
  * abnormal cardiac biomarkers (Abnormal high sensitivity TnT 5th generation levels (>9 ng/L: female, >14 ng/L: male) or abnormal age appropriate N terminal pro-brain natriuretic peptide, NT-proBNP (abnormal values: <50 years: >450 pg/ml; 50-75 years:>900 pg/ml; >75 years: >1800 pg/ml) or
  * abnormal echocardiogram (wall thickness > 12 mm) or
  * abnormal cardiac MRI (wall thickness > 12 mm or extracellular volume > 0.35) OR
* Diagnosis of transthyretin cardiac amyloidosis by standard criteria

  * endomyocardial biopsy followed by typing of the transthyretin amyloidosis using immunohistochemistry or immunogold assay with confirmation by Mass spectroscopy as needed
  * extracardiac biopsy with typical cardiac imaging findings, or
  * grade 2 or grade 3 myocardial uptake of technetium-99m pyrophosphate (PYP) if AL amyloidosis is excluded

Exclusion Criteria:

* Hemodynamic instability
* Severe claustrophobia despite use of sedatives
* Decompensated heart failure (unable to lie flat for 1 hour)
* Concomitant non-ischemic non-amyloid heart disease (valvular heart disease or dilated cardiomyopathy)
* Severe valve stenosis or regurgitation in the aortic, mitral or tricuspid valves, including prior valve replacement
* Severe pulmonary artery hypertension
* Severe lung disease
* Known obstructive epicardial coronary artery disease with stenosis > 50% in any single territory
* Prior cardiac surgery
* Regional wall motion abnormality on echocardiogram
* Left ventricular ejection fraction < 40%
* Pregnant state
* Documented allergy to N-13 ammonia or Definity
* Contraindications to DEFINITY® (Perflutren Lipid Microsphere) Injectable Suspension:

  o Patients with known or suspected Right-to-left, bi-directional, or transient right-to-left cardiac shunts, Hypersensitivity to perflutren
* Contraindications or challenges to sonotherapy

  * Severe electrolyte abnormalities
  * QTc prolongation (values are greater than 450 milliseconds in males and greater than 470 milliseconds in females)
  * BMI > 35 kg/m2
  * Documented intracardiac thrombus
  * Atrial fibrillation not on anticoagulation
  * Prior history of stroke
* Any other reason determined by the investigator that makes a subject a poor candidate for ultrasound therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial Blood Flow | 1 day
  N-13 ammonia or Rubidium-82 PET based measure of myocardial blood flow in ml/gm/min
Systolic Function | 1 day
  Global Longitudinal Strain by echocardiography
Diastolic Function | 1 day
  Echo measured mitral e' velocity

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Dorbala, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IRD